CLINICAL TRIAL: NCT01816958
Title: Treatment of Thalamocortical Dysrhythmia Using External Neuromodulation to Facilitate the Therapeutic Effect of Ketamine.
Brief Title: Neuromodulation to Facilitate the Effect of Ketamine
Acronym: TMS/ketamine
Status: Completed | Type: Observational
Sponsor: The Neuroscience Center, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 12_1293
Record Dates: First submitted 2013-03-11; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Depression; Chronic Pain; Substance Abuse
Keywords: thalamocortical dysrhythmia; transcranial magnetic stimulation (TMS); transcranial Electrical Stimulation (tES); (N-methyl-D-aspartate) NMDA-R antagonist; ketamine infusion; neuromodulation; synergistic effect; remission
MeSH Terms: conditions — Depression; Chronic Pain; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic depression and/or pain: co-administration of TMS and infused ketamine for patients with chronic pain of psyche and/or soma
  Interventions: Other: co-administration of TMS and infused ketamine

INTERVENTIONS:
Other: co-administration of TMS and infused ketamine — co-administration of TMS and infused ketamine

SUMMARY:
application of external neuromodulation along with ketamine infusion.

DETAILED DESCRIPTION:
apply TMS concurrent with ketamine infusion in order to increase the likliehood & strength of therapeutic benefit

ELIGIBILITY:
Inclusion Criteria:

* chronically ill,
* treatment-resistant

Exclusion Criteria:

* active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients within my own clinic, suffering with chronic emotional and/or somatic pain
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Function in DSM-4R | up to 3 years
  treat in order to cause remission of disability

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Devore Best, M.D., Principal Investigator — The Neuroscience Center
Locations (1):
- The Neuroscience Center, Deerfield, Illinois, United States